CLINICAL TRIAL: NCT04347382
Title: The Role of Honey and Nigella Sativa in the Management of COVID-19; A Randomized Controlled, Open-label, Add-on Trial in Pakistan
Brief Title: Honey & Nigella Sativa Trial Against COVID-19
Acronym: HNS-COVID-PK
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sohaib Ashraf (Other)
Responsible Party: Sponsor-Investigator, Sohaib Ashraf, Post-Graduate Resident Cardiology, Sheikh Zayed Federal Postgraduate Medical Institute
Organization: Sheikh Zayed Federal Postgraduate Medical Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SZMC/IRB/Internal/0026/2020; IRB/2020/658/SIMS (Other: Services Institute of Medical Sciences, Services Hospital, Lahore, Pakistan)
Record Dates: First submitted 2020-04-11; First posted 2020-04-15 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Coronavirus Infection; Sars-CoV2
Keywords: SARS-CoV-2; COVID-19; Coronavirus; Honey; Nigella Sativa; Black Cummin; Herbal Medicine
MeSH Terms: conditions — Coronavirus Infections; COVID-19 | interventions — Honey

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nigella Sativa & Honey Group (Experimental): Drug: Nigella Sativa seed Powder 80 mg/Kg/day grinded in capsule upto a max of 14 days) Drug: Natural Honey 1gm/kg/day orally upto a max of 14 days)
  along with standard medical care
  Interventions: Drug: Honey; Drug: Nigella Sativa / Black Cumin
- Standard Medical Care (Placebo Comparator): Standard supportive medical care prescribed by treating physician, Lahore which includes standard symptomatic care along with use of antibacterial or antiviral (if advised by pulmonologist or infectious disease specialist)
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Honey — 1gm/Kg/Day
  Arms: Nigella Sativa & Honey Group
Drug: Nigella Sativa / Black Cumin — 80mg/Kg/day
  Arms: Nigella Sativa & Honey Group
Drug: Placebos — Empty capsule with 250ml of distilled water
  Arms: Standard Medical Care

SUMMARY:
To evaluate the effectiveness of Nigella Sativa and honey stirred in 250 ml of distilled water 12 hourly till patient becomes asymptomatic or a maximum of 14 days with standard hospital care versus standard hospital care alone with placebo capsule and 250 ml water, in clearing the COVID-19 nucleic acid from throat and nasal swab, lowering disease detrimental effects on HRCT chest/X-ray and severity of symptoms along with duration of hospital stay till day 14th day of follow up and 30 days mortality (primary outcomes).

DETAILED DESCRIPTION:
This cohort, adaptive, randomized, double armed group, controlled, Investigator Initiated interventional study is designed to demonstrate the superiority of a combination of black cumin with honey over standard care in SARS-CoV-2 (COVID-19) infected patients who consent to randomization following a new diagnosis in Pakistan with an SSC-2 score of > 5 with positive RT-PCR of COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed SARS-CoV-2 (COVID-19) infection by a positive test result with SSC-2 score> 5
* Patients admitted in Corona centers

Exclusion Criteria:

* Participants not giving consent.
* Pregnant and lactating females.
* History of allergy to any drug being administered in this study
* Severely terminally ill patients
* Patients on Nil Per Oral

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2020-04-30 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Days required to get a positive COVID-19 PCR to negative | upto max 14 days
Severity of symptoms progression | upto max 14 days
  Clinically disease progression will be evaluated depending upon the severity of symptoms being classified as mild, moderate and severe.
Duration of Hospital Saty | upto max 14 day
  Duration of hospital stay would be categorized as the number of days the patient stayed in the ward during treatment. The date of admission and date of discharge would give us total duration of stay.
30 day mortality | 30 days
  30 days mortality rate in each arm
Clinical Grade Status | 0, 4, 6, 8, 10 and 12 day
  grade 1 (not hospitalized, no evidence of infection and resumption of normal activities), grade 2 (not hospitalized, but unable to resume normal activities), grade 3 (hospitalized, not requiring supplemental oxygen), grade 4 (hospitalized, requiring supplemental oxygen), grade 5 (hospitalized, requiring nasal high-flow oxygen therapy and/or noninvasive mechanical ventilation), grade 6 (hospitalized, requiring ECMO and/or invasive mechanical ventilation) and grade 7 (death).
Fever | 13 days
  Degree of fever

SECONDARY OUTCOMES:
Oxygen Saturation at room air | upto max of 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Shoaib Ashraf, PhD, Study Director — Massachusetts General Hospital, Harvard Medical School, USA; Muhammad Ashraf, DVM, PhD, Study Chair — University Of Veterinary & Animal Sciences, Lahore; Sohaib Ashraf, MBBS, Principal Investigator — Federal Post-Graduate Medical Institute, Lahore; Muhammad Ahmad Imran, MBBS, Principal Investigator — Shaikh Zayed Hospital, Lahore; Ayesha Hamayun, MBBS, PhD, Principal Investigator — Shaikh Khalifa Bin Zayed Al-Nahyan Medical & Dental College, Lahore
Locations (2):
- Pakistan (2):
  - Federal Post-Graduate Medical Institute, Shaikh Zayed Hospital, Lahore, Punjab Province
  - Services Institute of Medical Sciences, Services Hospital, Lahore, Punjab Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ulasli M, Gurses SA, Bayraktar R, Yumrutas O, Oztuzcu S, Igci M, Igci YZ, Cakmak EA, Arslan A. The effects of Nigella sativa (Ns), Anthemis hyalina (Ah) and Citrus sinensis (Cs) extracts on the replication of coronavirus and the expression of TRP genes family. Mol Biol Rep. 2014 Mar;41(3):1703-11. doi: 10.1007/s11033-014-3019-7. Epub 2014 Jan 12. PMID 24413991
- [Background] Oyero OG, Toyama M, Mitsuhiro N, Onifade AA, Hidaka A, Okamoto M, Baba M. SELECTIVE INHIBITION OF HEPATITIS C VIRUS REPLICATION BY ALPHA-ZAM, A NIGELLA SATIVA SEED FORMULATION. Afr J Tradit Complement Altern Med. 2016 Sep 29;13(6):144-148. doi: 10.21010/ajtcam.v13i6.20. eCollection 2016. PMID 28480371
- [Background] Khan SU, Anjum SI, Rahman K, Ansari MJ, Khan WU, Kamal S, Khattak B, Muhammad A, Khan HU. Honey: Single food stuff comprises many drugs. Saudi J Biol Sci. 2018 Feb;25(2):320-325. doi: 10.1016/j.sjbs.2017.08.004. Epub 2017 Aug 16. PMID 29472785
- [Background] Forouzanfar F, Bazzaz BS, Hosseinzadeh H. Black cumin (Nigella sativa) and its constituent (thymoquinone): a review on antimicrobial effects. Iran J Basic Med Sci. 2014 Dec;17(12):929-38. PMID 25859296
- [Derived] Ashraf S, Ashraf S, Ashraf M, Imran MA, Kalsoom L, Siddiqui UN, Farooq I, Akmal R, Akram MK, Ashraf S, Ghufran M, Majeed N, Habib Z, Rafique S, -Abdin ZU, Arshad S, Shahab MS, Ahmad S, Zheng H, Mirza AR, Zulfiqar S, Anwar MI, Humayun A, Mahmud T, Saboor QA, Ahmad A, Ashraf M, Izhar M; DOCTORS LOUNGE consortium. Honey and Nigella sativa against COVID-19 in Pakistan (HNS-COVID-PK): A multicenter placebo-controlled randomized clinical trial. Phytother Res. 2023 Feb;37(2):627-644. doi: 10.1002/ptr.7640. Epub 2022 Nov 24. PMID 36420866